CLINICAL TRIAL: NCT06228820
Title: Aspirin Resistance in Trinidad: The ART Pilot Study.
Brief Title: Aspirin Resistance in Trinidad.
Acronym: ART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Naveen Seecheran, Principal Investigator, The University of The West Indies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEC1153/06/19
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Platelet Dysfunction Due to Drugs
Keywords: Aspirin
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Healthy patients will then undergo at least a 2-week course of 81mg of Bayer Aspirin per oral daily, followed by platelet function testing. The patients will then undergo a washout period of 2 weeks, followed by another 2-week course of 81mg Vazalore Aspirin per oral daily, followed by a second round of platelet function testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aspirin Arm (Experimental): Healthy patients will then undergo at least a 2-week course of 81mg of Bayer Aspirin per oral daily, followed by platelet function testing. The patients will then undergo a washout period of 2 weeks, followed by another 2-week course of 81mg Vazalore Aspirin per oral daily, followed by a second round of platelet function testing.
  Interventions: Drug: Aspirin 81Mg Ec Tab

INTERVENTIONS:
Drug: Aspirin 81Mg Ec Tab — Healthy patients will then undergo at least a 2-week course of 81mg of Bayer Aspirin per oral daily, followed by platelet function testing. The patients will then undergo a washout period of 2 weeks, followed by another 2-week course of 81mg Vazalore Aspirin per oral daily, followed by a second round of platelet function testing.

SUMMARY:
Aspirin's beneficial effect is mediated via the inhibition of arachidonic acid (AA) activation of platelets. It is detected by demonstrating a decrease in platelet function and/or a decrease in prostaglandin metabolites. Besides inhibiting the formation of thromboxane A2 from arachidonic acid, Aspirin has a host of platelet-independent effects that complement its platelet-inhibitory effects.

The phenomenon of "Aspirin resistance" is based on the observation of clinical events in some patients taking Aspirin and/or a diminished platelet aggregation inhibitory response to Aspirin therapy. It has been suggested that many individuals taking Aspirin have become resistant to this drug. Unfortunately, laboratory assays used to monitor the efficacy of Aspirin are far from accurate, and the results are not reproducible. Multiple studies demonstrate non-compliance using repeat testing for platelet inhibition in patients with an initial inadequate response to Aspirin. When the test is repeated under the condition that the ingestion of the test Aspirin is assured, the patients' platelets are inhibited. Patients with an inadequate Aspirin response have an increased likelihood of subsequent vascular events.

DETAILED DESCRIPTION:
Aspirin is a wonder drug used for over 100 years for its analgesic and antipyretic effects. It is an inexpensive, readily available medication that reduces the risk of subsequent vascular disease by about 25% in patients with known occlusive vascular disease. For the past three decades, it has increasingly been used to prevent primary and secondary cardiovascular events.

Aspirin's beneficial effect is mediated via the inhibition of arachidonic acid (AA) activation of platelets. It is detected by demonstrating a decrease in platelet function and/or a decrease in prostaglandin metabolites. Besides inhibiting the formation of thromboxane A2 from arachidonic acid, Aspirin has a host of platelet-independent effects that complement its platelet-inhibitory effects.

The phenomenon of "Aspirin resistance" is based on the observation of clinical events in some patients taking Aspirin and/or a diminished platelet aggregation inhibitory response to Aspirin therapy. It has been suggested that many individuals taking Aspirin have become resistant to this drug. Unfortunately, laboratory assays used to monitor the efficacy of Aspirin are far from accurate, and the results are not reproducible. Multiple studies demonstrate non-compliance using repeat testing for platelet inhibition in patients with an initial inadequate response to Aspirin. When the test is repeated under the condition that the ingestion of the test Aspirin is assured, the patients' platelets are inhibited. Patients with an inadequate Aspirin response have an increased likelihood of subsequent vascular events.

The POINT pilot study introduced the preliminary observation that the estimated prevalence of HPR is considerably higher within the heterogeneous population in Trinidad at 50% compared with predominantly Caucasian studies. Furthermore, the HPR is significantly higher in South Asians (Indo-Trinidadians) (>60% of patients), which has severe clinical repercussions considering the cardiovascular disease pandemic. Clopidogrel may not be a satisfactory or optimal antiplatelet agent in this subgroup. Therefore, another more potent antiplatelet, such as ticagrelor, should be used instead.

Patients generally displayed a limited level of cardiovascular medication adherence, which is likely to translate into a higher rate of cardiovascular events with their potentially devastating sequelae.

We postulate that there is a high level of Aspirin resistance in Trinidad and Tobago.

ELIGIBILITY:
Inclusion Criteria:

1. between 18 and 74 years of age,
2. healthy with no overt medical conditions,
3. not on any physician-prescribed medications or complementary/alternative therapies,

Exclusion Criteria:

1. presence of active internal bleeding or history of bleeding diathesis or clinical findings associated with an increased risk of bleeding,
2. history of ischemic or hemorrhagic stroke, transient ischemic attack, intracranial neoplasm, arteriovenous malformation, or aneurysm,
3. clinical and/or hemodynamic instability,
4. within 1 month of placement of a bare metal stent,
5. within 30 days of coronary artery bypass graft surgery or PCI without a stent placed,
6. planned coronary revascularization,
7. treatment with fibrin-specific fibrinolytic therapy <24 h or non-fibrin-specific fibrinolytic therapy <48 h,
8. use of an oral anticoagulation agent or international normalized ratio >1.5,
9. body weight <60 kg,
10. age >75 years,
11. hemoglobin <10 g/dL,
12. platelet count <100×106/μL,
13. creatinine >2 mg/dL,
14. hepatic enzymes >2.5 times the upper limit of normal,
15. pregnancy and/or lactation,
16. the patient is on any other antithrombotic therapies such as ticagrelor, dabigatran, rivaroxaban and apixaban

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders are included.
Enrollment: 48 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Aspirin Resistance Unit | 2-weeks
  VerifyNow Aspirin assay is a qualitative test to aid in detecting platelet dysfunction due to Aspirin ingestion in whole blood for the point-of-care or laboratory setting. The assay incorporates the agonist arachidonic acid to activate platelets, and it measures platelet function based on the ability of activated platelets to bind to fibrinogen. Fibrinogen-coated microparticles aggregate in whole blood in proportion to the number of activated platelet GP IIb/IIIa receptors. If Aspirin has produced the expected antiplatelet effect, such aggregation will be reduced. The VerifyNow Aspirin assay reports the extent of platelet aggregation as Aspirin reaction units (ARUs). Given an ARU range of 350-700, ARU values less than 550 are consistent with Aspirin-induced inhibition of platelet function. In contrast, values greater than or equal to 550 ARUs are not compatible with Aspirin-induced inhibition.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of the West Indies, Saint Augustine, North, Trinidad and Tobago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seecheran N, McCallum P, Grimaldos K, Ramcharan P, Kawall J, Katwaroo A, Seecheran V, Jagdeo CL, Rafeeq S, Seecheran R, Quert AL, Ali N, Peram L, Khan S, Ali F, Motilal S, Bhagwandass N, Giddings S, Ramlackhansingh A, Sandy S. Pharmacodynamic Comparison of Two Aspirin Formulations in the Caribbean: The ARC Study. Cardiol Ther. 2024 Sep;13(3):593-602. doi: 10.1007/s40119-024-00373-6. Epub 2024 Jul 15. PMID 39008026